CLINICAL TRIAL: NCT05731011
Title: Effects of Physical Therapy on Oxidative Stress
Brief Title: Effects of Physical Therapy on Oxidative Stress in Female Patients With Gonarthrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, mustafa gulsen, assocc.prof., Baskent University
Other Study IDs: KA22/363
Record Dates: First submitted 2023-02-06; First posted 2023-02-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Gonarthrosis; Antioxidative Stress
Keywords: gonarthrosis; antioxidative stress
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Oxidative Stress; Electric Stimulation Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Other: antioxidative stress — blood interventions
  Other Names: electrotherapy
Device: electrotherapy — hotpack,Tens, ultrasound

SUMMARY:
This study aimed to investigate the production of reactive oxygen derivatives (ROS) and reactive nitrogen derivatives (RNT) in female patients with knee OA, and their effects on oxidative stress by evaluating before and after physical therapy in female patients with gonarthrosis who have Kellegren-Lawrence Staging Scale Stage II and III. aimed. To this study; All female cases over the age of 40 who applied to Başkent University Ankara Hospital and were diagnosed with knee OA by a specialist doctor will be included.

Method After the cases participating in the study were checked by a specialist physician, the cases that did not prevent them from being included in the study; It will be graded according to the Kellegren-Lawrence Staging Scale. Stage II and III cases will be included in the study. Sociodemographic characteristics of the patients will be recorded before the treatment. 10 sessions of physical therapy program will be applied to the patients. Treatment program 20 minutes Hot pack (HP), 60-100 Hz frequency range, 60 pulse duration and 20 minutes of conventional TENS (Enraf-NoniusBDelftechpark 39, 2600 AV, Delft, The Netherlands) with the patient comfortable feeling and 10 minutes continuous around the knee A home exercise program will be given with ultrasound (Enraf-Nonius-B Delftechpark 39; 1-MHz; 1.5 watts/cm2) to strengthen the muscles around the knees. Those with acute inflammation of the knee joint, those who underwent surgery in the knee joint for any reason or any trauma to the lower extremity, those with a history of uncontrollable high blood pressure, any neurological or vestibular problems, those who have used steroid injections in the last two months, and any For this reason, patients with systemic diseases that will affect the study will be excluded from the study.

Staging criteria according to Kellegren-Lawrence Staging Scale; Stage 0: Normal Stage 1: Possible osteophyte Stage 2: Definite osteophyte, suspected narrowing of joint space Stage 3: Moderate osteophyte, definite narrowing Stage 4: Extensive osteophyte, marked narrowing, sclerosis (Kellegren and Lawrence, 1957).

Biochemical analyzes:

To this study; Blood samples will be taken before and after treatment from a female patient over 40 years old who was diagnosed with knee OA at Başkent University Ankara Hospital. Total antioxidant level (TAS): It will be determined by an automatic measurement method based on the fact that the characteristic color formed by the 2,2'azino-bis (3-ethylbenz-thiazoline-6-sulfonic acid) (ABTS) radical is brightened by the antioxidants in the sample added to the medium (Erel, 2004). Results will be given in mmol Trolox eqivalen/L.

Total oxidant level (TOS): will be determined by automatic measurement method (Erel, 2005). The oxidants in the sample have the task of converting the ferrous ion complex to a ferric ion. Ferric ion (Fe3+) formed by oxidation of iron (Fe2+) to its more stable form (Fe2O3) creates color with xylenol orange in acidic environment. The intensity of the color measured spectrophotometrically is related to the total amount of oxidant molecules present in the sample. The measurement is calibrated with hydrogen peroxide (H2O2) and the results will be given as micromolar H2O2 equivalent per liter (µmol H2O2 equiv./L) (Sydow, 1985).

Nitric oxide (NO): Serum nitric oxide concentration (Mirand et al, 2001) will be measured in a spectrophotometer according to the method (PowerWawe XS, BioTek, USA). Serum samples will be deproteinized with 10% zinc sulfate. In this method, nitrate was converted to nitrite with Vanadium (III) chloride. It is based on the measurement of the complex diazonium compound as a result of the reaction of nitrite and sulfanilamide N-(1-Naphthy) ethylene diamine dihydrochloride in an acidic medium.

High-density lipoprotein (HDL): It will be run in an autoanalyzer using the Biotrol trademark kit and given in mg/dl. The results will be recorded for each individual on the information sheet.

ELIGIBILITY:
Inclusion Criteria:

* Cases with Grade II and III Study Grades according to the Kellgren-Lawrence Staging Scale
* women over 40

Exclusion Criteria:

* Patients with acute inflammation of the knee joint,
* undergoing surgery in the knee joint for any reason or any trauma to the lower extremity,
* a history of uncontrollable high blood pressure,
* any neurological or vestibular problem,
* use of steroid injections in the last two months,
* any cases with systemic disease that may affect the study

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All female cases over 40 years old diagnosed with knee OA
Study Population: After the cases participating in the study were checked by a specialist physician, the cases that did not prevent them from being included in the study; It will be graded according to the Kellegren-Lawrence Staging Scale. Cases with Stage II and III will be included in the study.
Sampling Method: Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2023-08-25 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
antioxidant level | 2 months
  Blood samples will be taken before and after treatment. Total antioxidant level (TAS): It will be determined by an automatic measurement method based on the fact that the characteristic color formed by the 2,2'azino-bis (3-ethylbenz-thiazoline-6-sulfonic acid) (ABTS) radical is brightened by the antioxidants in the sample added to the medium (Erel, 2004). Results will be given in mmol Trolox eqivalen/L.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Gulsen, Principal Investigator — Baskent University
Locations (1):
- The Effects of Physical Therapy on Oxidative Stress in Female Patients With Gonarthrosis, Ankara, Turkey (Türkiye)